CLINICAL TRIAL: NCT00726622
Title: A Phase III Prospective Randomized Trial Comparing Laparoscopic-Assisted Resection Versus Open Resection for Rectal Cancer
Brief Title: Laparoscopic-Assisted Resection or Open Resection in Treating Patients With Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z6051; ACOSOG-Z6051; U10CA076001 (NIH); NCI-2009-00350 (Other: NCI Clinical Trial Reporting Office); CDR0000601816 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2008-07-31; First posted 2008-08-01 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Open laparotomy and rectal resection (Active Comparator): Patients undergo open laparotomy and rectal resection. The standard form of surgery is open laparotomy rectal resection. During open laparotomy, the surgeon makes a large incision or cut in the abdomen, and goes in through that cut to remove the tumor and lymph nodes from the rectum.
  Interventions: Procedure: Open laparotomy and rectal resection
- Arm 2: Laparoscopic-assisted rectal resection (Experimental): Patients undergo laparoscopic-assisted rectal resection. Laparoscopic-assisted rectal resection is performed using small instruments on long handles introduced into the abdomen through small ports called trocars in 3 - 6 positions on the abdomen through incisions measuring 5 -10 mm, under the guidance of a video camera. The abdominal wall is held up with carbon dioxide under pressure. The piece of bowel or intestine is removed through another incision (about 8 centimeters), and the ends of the intestine are reconnected to provide normal bowel function.
  Interventions: Procedure: Laparoscopic-assisted rectal resection

INTERVENTIONS:
Procedure: Open laparotomy and rectal resection — Patients undergo open laparotomy and rectal resection.
  Arms: Arm 1: Open laparotomy and rectal resection
Procedure: Laparoscopic-assisted rectal resection — Patients undergo laparoscopic-assisted rectal resection.
  Arms: Arm 2: Laparoscopic-assisted rectal resection

SUMMARY:
This study is being done to compare two types of surgery currently used for rectal cancer. The two types of surgery are laparoscopic-assisted rectal resection and open laparotomy rectal resection. Although laparoscopic-assisted rectal resection is being used for rectal cancer in some medical centers, the effectiveness of this type of surgery compared to open surgery is unknown. The study will compare the safety and effectiveness of the surgeries, recovery from surgery in the hospital, overall recovery from surgery and cancer outcome.

DETAILED DESCRIPTION:
This is a multicenter study. Patients eligible for this trial will have completed 5FU based neoadjuvant chemotherapy/radiation therapy per the institution's standard of care or IRB approved clinical trial. Patients may be registered/randomized anytime after completion of neoadjuvant therapy, but surgery must occur within 4-12 weeks (28-84 days) after completion of neoadjuvant therapy. Patients are stratified according to the site of the primary tumor (high, middle or low rectum), registering surgeon, and planned operative procedure (low anterior resection or abdominal perineal resection). Patients are randomized to 1 of 2 treatment arms. Please see the arms section for more details. The primary and secondary objectives are listed below.

Primary Objective:

To test the hypothesis that laparoscopic-assisted resection for rectal cancer is not inferior to open rectal resection, based on a composite primary endpoint of oncologic factors which are indicative of a safe and feasible operation.

Secondary Objectives:

1. To assess patient-related benefit of laparoscopic-assisted resection for rectal cancer vs.

   open rectal resection (blood loss, length of stay, pain medicine utilization)
2. To assess disease free survival and local pelvic recurrence at two years.
3. To assess quality of life, sexual function, bowel and stoma function at scheduled time points throughout the trial.

Patients will be evaluated after surgery to determine the need for subsequent care based on the final pathology. Patients should not start treatment on any other investigative trial involving intervention or invasive diagnostic procedures ≤ 30 days following surgery to enable a complete evaluation of post-operative adverse events and complications occurring within 30 days of surgery. Patients are followed periodically for up to 5 years post surgery.

ELIGIBILITY:
Eligibility Criteria:

1. Histologic diagnosis of adenocarcinoma of the rectum (≤ 12 cm from the anal verge)
2. T3, N0, M0, T1-3, N1-2, M0 disease as determined by pre-neoadjuvant therapy CT scans and pelvic MRI or transrectal ultrasound. Patients with T4 disease are not eligible.
3. Completion of pre-operative 5FU based chemotherapy and/or radiation therapy. Capecitabine may be substituted for 5FU.
4. Age ≥ 18 years
5. ECOG (Zubrod) Performance Status ≤ 2
6. Body Mass Index (BMI) ≤ 34
7. No evidence of conditions that would preclude use of a laparoscopic approach (eg, multiple previous major laparotomies, severe adhesions)
8. No systemic disease (cardiovascular, renal, hepatic) that would preclude surgery. No other severe incapacitating disease:

   * ASA IV: A patient with severe systemic disease that is a constant threat to life. OR
   * ASA V: A moribund patient who is not expected to survive without the operation.
9. No concurrent or previous invasive pelvic malignancy (cervical, uterine and rectal) within five years prior to registration
10. No history of psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

NOTE: Incompetent patients are not eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W. Fleshman, MD, Study Chair — Baylor Health
Locations (37):
- United States (35):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Clarian North Medical Center, Carmel, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Kendrick Regional Center for Colon and Rectal Care - Mooresville, Mooresville, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Blodgett Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Boone Hospital Center, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Overlook Hospital, Summit, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - INTEGRIS Cancer Institute of Oklahoma - Proton Campus, Oklahoma City, Oklahoma
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Forbes Regional Hospital, Monroeville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (2):
  - St. Paul's Hospital at Providence Health Care - Vancouver, Vancouver, British Columbia
  - St. Joseph's Hospital - Charlton Campus, Hamilton, Ontario

REFERENCES:
- [Derived] Fleshman J, Branda M, Sargent DJ, Boller AM, George V, Abbas M, Peters WR Jr, Maun D, Chang G, Herline A, Fichera A, Mutch M, Wexner S, Whiteford M, Marks J, Birnbaum E, Margolin D, Larson D, Marcello P, Posner M, Read T, Monson J, Wren SM, Pisters PW, Nelson H. Effect of Laparoscopic-Assisted Resection vs Open Resection of Stage II or III Rectal Cancer on Pathologic Outcomes: The ACOSOG Z6051 Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1346-55. doi: 10.1001/jama.2015.10529. PMID 26441179
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Started | 243 | 243
Completed | 225 | 240
Not Completed | 18 | 3
Not completed — Withdrawal by Subject | 16 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Metastasis | 2 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were randomized to a treatment arm were available for baseline characteristics. Four patients from Arm 1: Open laparotomy and rectal resection and one patient from Arm 2: Laparoscopic-assisted rectal resection are not shown because of patient refusal or improper consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection | Total
Number analyzed (Participants) | 239 | 242 | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.1) | 57.7 (11.5) | 57.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 86 | 167
  Male | 158 | 156 | 314
Region of Enrollment [Number; unit: participants]
  United States | 239 | 242 | 481

OUTCOME MEASURES:

1. Primary Outcome: Comparing Laparoscopic-assisted Resection to Open Rectal Resection for Rectal Cancer as Measured by the Percentage of Patients With Successful Resection Based on Pathological Evaluation.
Description: The primary endpoint will be a composite endpoint of oncologic factors which are indicative of an adequate surgical resection based on pathologic evaluation.
  Primary endpoint parameters:
  * Circumferential margin > 1 mm
  * Negative distal margin
  * Completeness of total mesorectal excision (TME) A complete TME is a rectal resection specimen that has an intact mesorectum and covering peritoneal envelope all the way to the level of rectal transection with no coning in of the mesorectum above the point of transection. The surface of the peritoneal covering should be smooth and shiny with no defects exposing the underlying fat.
  All three criteria must be met for a resection to be deemed adequate. Laparoscopic-assisted resection will be compared to Open rectal resection to determine if it is non-inferior.
Time Frame: At time of Surgery
Population: Of the 225 patients that received intervention as randomized in Arm 1: Open laparotomy and rectal resection, 3 patients were excluded from the analysis due to improper consent. All 240 patients from Arm 2 that received intervention as randomized were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Number analyzed (Participants) | 222 | 240
percentage of participants | 86.9 [82.5 to 91.4] | 81.7 [76.5 to 86.9]
Statistical Analysis 1: Comparison: Arm 1: Open Laparotomy and Rectal Resection vs Arm 2: Laparoscopic-assisted Rectal Resection; Test type: Non-Inferiority or Equivalence — Assuming a baseline rate of 90% oncologic success for the open resection arm, the sample size provided 80% power to declare non-inferiority if oncologic success rates were truly identical, using a 1-sided z score with α = .10 for falsely declaring non-inferiority when the true oncologic success rate for laparoscopic resection was 84%. Calculations were based on a 2-sample binomial non-inferiority calculation with a 90% success rate for the control group and a 6% non-inferiority margin; p = 0.41, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Completeness of Total Mesorectal Excision (Complete or Nearly Complete)
Description: Complete total mesorectal excision was defined as a rectal resection specimen having smooth surface of mesorectal fascia with all fat contained in the enveloping fascia to a level 5 cm below the tumor for tumor-specific total mesorectal excision for upper rectal cancer, or the entire mesorectal envelope present for low rectal cancer. Nearly complete was defined as a rectal resection specimen having the mesorectal envelope intact except for defects no more than 5 mm deep, with no loss of mesorectal fat.
  The percentage of patients with complete or nearly complete mesorectal excision was calculated along with the binomial 95% CI.
Time Frame: At time of surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Number analyzed (Participants) | 222 | 240
percentage of participants | 95.1 [92.2 to 97.9] | 92.1 [88.7 to 95.5]

3. Secondary Outcome: Negative Distal Resected Margin
Description: The percentage of patients with negative distal margin (>1 mm between the closest tumor to the cut edge of the tissue) was calculated along with binomial 95% confidence intervals.
Time Frame: At time of surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Number analyzed (Participants) | 222 | 240
percentage of participants | 98.2 [96.5 to 99.95] | 98.3 [96.7 to 99.95]

4. Secondary Outcome: Circumferential Margin > 1 mm
Description: The distance between the closest tumor to the cut edge of the tissue was measure post-resection. The percentage of patients with >1mm between the closest tumor to the cut edge of the tissue was calculated with a binomial 95% confidence interval.
Time Frame: At time of surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Number analyzed (Participants) | 222 | 240
percentage of participants | 92.3 [88.8 to 95.8] | 87.9 [83.8 to 92.0]

5. Secondary Outcome: Length of Stay
Description: The mean number of days required post-surgery to the when the patient was released from the hospital was calculated.
Time Frame: Two weeks post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Number analyzed (Participants) | 222 | 240
days | 7.0 (3.4) | 7.3 (5.4)

6. Secondary Outcome: Use of Pain Medication
Description: The number of days patients received parenteral narcotics post-surgery were counted.
Time Frame: Two weeks post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Number analyzed (Participants) | 222 | 240
days | 4.2 (2.8) | 4.2 (3.9)

7. Secondary Outcome: Operative Times
Description: Open to close operative time.
Time Frame: During surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Number analyzed (Participants) | 222 | 240
minutes | 220.6 (92.4) | 266.2 (101.9)

8. Secondary Outcome: Disease-free Survival
Time Frame: Up to 2 years post surgery
Reporting Status: Not Posted

9. Secondary Outcome: Local Pelvic Recurrence Rates
Time Frame: Up to 2 years post surgery
Reporting Status: Not Posted

10. Secondary Outcome: Overall Survival
Time Frame: Up to 5 years post surgery
Reporting Status: Not Posted

11. Secondary Outcome: Quality of Life and Sexual Function
Time Frame: Up to 5 years post surgery
Reporting Status: Not Posted

12. Secondary Outcome: Bowel Function
Time Frame: Up to 5 years post surgery
Reporting Status: Not Posted

13. Secondary Outcome: Bowel and Stoma Function
Time Frame: Up to 5 years post surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were collected after surgery and were collected up to 30 days after surgery.
Description: All patients that were randomized to a treatment arm were available for adverse event analysis. Four patients from Arm 1: Open laparotomy and rectal resection and one patient from Arm 2: Laparoscopic-assisted rectal resection are not shown because of patient refusal or improper consent. Therefore, this analysis is based on 239 patients on Arm 1 and 242 Patients on Arm 2.
Arm/Group | Arm 1: Open Laparotomy and Rectal Resection | Arm 2: Laparoscopic-assisted Rectal Resection
Serious Adverse Events (participants affected / at risk) | 11/239 | 10/242
Other Adverse Events (participants affected / at risk) | 201/239 | 207/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Open Laparotomy and Rectal Resection (N=239) | Arm 2: Laparoscopic-assisted Rectal Resection (N=242)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (2)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Intraoperative complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Intraoperative gastrointestinal injury - Pancreas (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
INR increased (Investigations) | 1 (1) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Open Laparotomy and Rectal Resection (N=239) | Arm 2: Laparoscopic-assisted Rectal Resection (N=242)
Blood disorder (Blood and lymphatic system disorders) | 3 (13) | 3 (6)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 33 (51) | 31 (46)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 5 (9) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (4) | 1 (2)
Cardiac pain (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 4 (5) | 4 (4)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 7 (7) | 8 (8)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Endocrine disorder (Endocrine disorders) | 2 (3) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 14 (19) | 12 (16)
Abdominal pain (Gastrointestinal disorders) | 32 (57) | 45 (72)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Anal pain (Gastrointestinal disorders) | 4 (4) | 5 (7)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Cecal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 18 (23) | 18 (20)
Diarrhea (Gastrointestinal disorders) | 43 (87) | 44 (74)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 4 (4) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (2)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 64 (117) | 53 (101)
Flatulence (Gastrointestinal disorders) | 6 (6) | 5 (7)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 24 (37) | 31 (43)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 5 (7) | 1 (1)
Ileal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 39 (47) | 35 (40)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 43 (70) | 54 (88)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Proctoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 16 (28) | 8 (12)
Rectal hemorrhage (Gastrointestinal disorders) | 5 (6) | 8 (8)
Rectal pain (Gastrointestinal disorders) | 79 (149) | 85 (153)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal stenosis (Gastrointestinal disorders) | 12 (21) | 14 (28)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 24 (28) | 17 (19)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 22 (28) | 25 (36)
Chest pain (General disorders) | 6 (7) | 4 (4)
Chills (General disorders) | 4 (4) | 4 (4)
Disease progression (General disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 10 (13) | 11 (12)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 49 (114) | 48 (73)
Fever (General disorders) | 19 (23) | 27 (34)
Flu-like symptoms (General disorders) | 1 (1) | 1 (1)
Gait abnormal (General disorders) | 0 (0) | 2 (3)
General symptom (General disorders) | 3 (3) | 4 (4)
Localized edema (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 20 (31) | 19 (27)
Visceral edema (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 6 (7) | 3 (4)
Anal infection (Infections and infestations) | 3 (3) | 2 (2)
Anorectal infection (Infections and infestations) | 5 (5) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 3 (3) | 4 (6)
Device related infection (Infections and infestations) | 0 (0) | 1 (2)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Ileal infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 13 (26) | 15 (23)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 2 (3) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 5 (7) | 3 (3)
Peritoneal infection (Infections and infestations) | 3 (4) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 6 (7) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 3 (5) | 5 (5)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 17 (21) | 16 (20)
Wound infection (Infections and infestations) | 17 (23) | 17 (21)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Intestinal stoma leak (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Intestinal stoma obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Intraoperative complications (Injury, poisoning and procedural complications) | 21 (29) | 14 (28)
Intraoperative neurological injury - NERVES: CN IX (glossopharyngeal) motor pharynx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Large intestinal anastomotic leak (Injury, poisoning and procedural complications) | 2 (4) | 3 (3)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 5 (5) | 5 (6)
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 5 (6) | 3 (3)
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 8 (11) | 5 (6)
Seroma (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureteric anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urethral anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Urostomy leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 26 (37) | 18 (34)
Alanine aminotransferase increased (Investigations) | 4 (8) | 3 (6)
Alkaline phosphatase increased (Investigations) | 4 (9) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 4 (7) | 4 (7)
Bilirubin increased (Investigations) | 2 (2) | 2 (2)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Coagulopathy (Investigations) | 2 (2) | 3 (3)
Creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 7 (8) | 7 (8)
INR increased (Investigations) | 1 (2) | 2 (3)
Laboratory test abnormal (Investigations) | 9 (17) | 6 (10)
Leukocyte count decreased (Investigations) | 5 (6) | 13 (18)
Lymphocyte count decreased (Investigations) | 2 (2) | 6 (8)
Neutrophil count decreased (Investigations) | 4 (4) | 7 (8)
Platelet count decreased (Investigations) | 10 (15) | 9 (12)
Serum cholesterol increased (Investigations) | 1 (1) | 1 (1)
Weight gain (Investigations) | 2 (4) | 1 (1)
Weight loss (Investigations) | 16 (27) | 13 (21)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 22 (29) | 14 (20)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 11 (17) | 11 (23)
Dehydration (Metabolism and nutrition disorders) | 26 (32) | 14 (22)
Serum albumin decreased (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 9 (10) | 5 (6)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 6 (8) | 2 (3)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Serum potassium decreased (Metabolism and nutrition disorders) | 14 (18) | 11 (13)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 8 (9) | 6 (6)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (23) | 8 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (10)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6 (10) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (7) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9) | 7 (8)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 10 (12) | 8 (9)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (6) | 8 (9)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Myelitis (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neurological disorder NOS (Nervous system disorders) | 4 (4) | 5 (10)
Peripheral motor neuropathy (Nervous system disorders) | 1 (5) | 5 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 35 (72) | 39 (83)
Radiculitis brachial (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 3 (3)
Taste alteration (Nervous system disorders) | 3 (3) | 2 (3)
Agitation (Psychiatric disorders) | 2 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 8 (11) | 4 (12)
Confusion (Psychiatric disorders) | 4 (4) | 4 (4)
Depression (Psychiatric disorders) | 10 (26) | 16 (30)
Insomnia (Psychiatric disorders) | 9 (16) | 12 (20)
Libido decreased (Psychiatric disorders) | 3 (4) | 1 (2)
Orgasm abnormal (Psychiatric disorders) | 50 (124) | 39 (95)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 2 (2) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 2 (4) | 2 (2)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 7 (7) | 5 (5)
Ureteric obstruction (Renal and urinary disorders) | 3 (5) | 2 (2)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (2) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 7 (8) | 7 (12)
Urinary incontinence (Renal and urinary disorders) | 4 (8) | 6 (6)
Urinary retention (Renal and urinary disorders) | 26 (43) | 40 (54)
Urine discoloration (Renal and urinary disorders) | 2 (2) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 8 (11) | 4 (4)
Vesical fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 3 (8) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 65 (177) | 64 (152)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 5 (11) | 11 (26)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal atresia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 3 (4)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vaginal stricture (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (12) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 11 (14)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (11) | 6 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 11 (15) | 5 (7)
Skin disorder (Skin and subcutaneous tissue disorders) | 12 (18) | 19 (29)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Sweating (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4)
Hematoma (Vascular disorders) | 6 (7) | 5 (5)
Hemorrhage (Vascular disorders) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 7 (9)
Hypotension (Vascular disorders) | 12 (13) | 8 (9)
Lymph leakage (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 10 (14) | 9 (10)
Vascular disorder (Vascular disorders) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes